CLINICAL TRIAL: NCT06029374
Title: Conservative Therapy of Fifth Metacarpal Neck Fractures - a Prospective Randomized Study Comparing Functional Treatment With Reposition and Finger Splinting
Brief Title: Therapy of Fifth Metacarpal Neck Fractures - Comparing Functional Treatment With Reposition and Finger Splinting
Acronym: BoxerFx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Paul L Hoppe, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1529/2023
Record Dates: First submitted 2023-08-26; First posted 2023-09-08 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Boxer's Fracture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Treatment (Active Comparator)
  Interventions: Procedure: Functional Treatment
- Forearm Cast and Finger Splint (Active Comparator)
  Interventions: Procedure: Forearm Cast and Finger Splint

INTERVENTIONS:
Procedure: Functional Treatment — Patients receiving buddy taping for fingers IV and V and an elastic bandage in terms of a functional treatment. Duration of bandage treatment is determined with 4 weeks.
  Arms: Functional Treatment
Procedure: Forearm Cast and Finger Splint — Patients receiving reduction of fractured finger and subsequent customization of a forearm cast with a finger splint. Duration of cast treatment is determined with 4 weeks.
  Arms: Forearm Cast and Finger Splint

SUMMARY:
The purpose of this prospective randomized controlled clinical trial is to evaluate if functional treatment leads to a better functional outcome than a forearm cast and a finger splint in patients with fifth metacarpal neck fracture.

DETAILED DESCRIPTION:
This study represents a prospective randomized clinical trial comparing two different conservative treatment options in patients with fifth metacarpal neck fracture.

Patients meeting the inclusion criteria will be enrolled in the present study provided they give their consent. Informed written consent will be obtained. Randomization will be performed according to the CONSORT Guidelines of Prospective Randomized Trials using the software "Randomizer" by the Medical University of Graz. Patients allocated to the control group will receive a forearm cast with a finger splint in terms of an immobilizing treatment, while patients in the study group will receive buddy taping for fingers IV and V and an elastic bandage in terms of a functional treatment. Both groups will receive the allocated bandage or splint for 4 weeks. The clinical outcome will be assessed 12 weeks after trauma.

ELIGIBILITY:
Inclusion Criteria:

* Fifth Metacarpal Neck Fractures
* Patient age between 18 and 70 years

Exclusion Criteria:

* Palmar angulation >50° in first lateral x-ray
* Pathologic fracture
* Intraarticular fracture
* Patients unable to consent
* Polytraumatized patients
* Pregnancy
* Compound fractures
* Multiple hand injuries
* Patients initially presenting more than 7 days after injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Brief Michigan-Hand-Outcome-Questionnaire | at 12 weeks
  patient-based standardised questionnaire (12 items, range 0-100, 100=ideal function, 0=poorest function)

SECONDARY OUTCOMES:
Loss/Gain of Reduction | at 12 weeks
  changes in palmar angulation of the fracture at end of treatment, compared to first x-ray (in degrees)
Treatment Failure | at 1, 2, 4 and 12 weeks
  Occurrence of indication for surgery (malrotation, palmar angulation >50°) after primary reposition

OTHER OUTCOMES:
Visual Analogue Scale (VAS) | at 0, 1, 2, 4 and 12 weeks
  Pain evaluation on a psychometric response scale (range 0-10, 0=no pain, 10=maximum pain)
Strength Measurement | at 4 and 12 weeks
  dynamometer-based strength evaluation
Range of Motion (ROM) Assessment | at 4 and 12 weeks
  goniometer-based ROM evaluation of hand and wrist
Delayed Bone Healing | at 12 weeks
  number of participants with bone non-union at end of study
Radiological Outcome | at 0, 1, 2, 4 and 12 weeks
  x-ray based outcome of fracture healing in terms of axial deviation (measured in degrees)
Radiological Outcome | at 0, 1, 2, 4 and 12 weeks
  x-ray based outcome of fracture healing in terms of length deviation and dislocation (measured in mm)
Quick DASH-Score | at 0, 1, 2, 4 and 12 weeks
  patient-based standardised questionnaire (11 items, range 0-100, 100=ideal function, 0=poorest function)
Brief Michigan-Hand-Outcome-Questionnaire | at 0, 1, 2 and 4 weeks
  patient-based standardised questionnaire (12 items, range 0-100, 100=ideal function, 0=poorest function)
Occurrence of Complications | at 0, 1, 2, 4 and 12 weeks
  occurence of complications due to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gerhild Thalhammer, M.D., Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna - Department of Orthopedics and Trauma-Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No